CLINICAL TRIAL: NCT04753476
Title: The Effect of Secretome of Hypoxia-Mesenchymal Stem Cells in Improving Survival of Severe Covid-19 Patients
Brief Title: Treatment of Severe COVID-19 Patients Using Secretome of Hypoxia-Mesenchymal Stem Cells in Indonesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cell and Cancer Research Indonesia (Network)
Collaborators: Provincial Government of Central Java, Indonesia (Unknown)
Responsible Party: Principal Investigator, Agung Putra, Assoc. Prof. Dr. dr. Agung Putra, M.Si. Med, Stem Cell and Cancer Research Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCR_Secretome
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Covid-19; Cytokine Storm
Keywords: secretome; mesenchymal stem cells; covid-19; hypoxia
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secretome-MSCs (n=24) (Experimental): This group will be given Covid-19 standard therapy with intramuscular Hypoxic S-MSC secretome
  Interventions: Biological: Injection of Secretome-MSCs; Drug: Standard treatment of Covid-19
- Control (n=24) (Other): This group will receive standard Covid-19 therapy with the best supportive care
  Interventions: Drug: Standard treatment of Covid-19

INTERVENTIONS:
Biological: Injection of Secretome-MSCs — Injection of Hypoxic Secretome-MSCs intramuscular (deltoideus) :
  Day 1: 1 cc every 12 hours
  Day 2: 1 cc every 12 hours
  Day 3: 1 cc every 12 hours
  Arms: Secretome-MSCs (n=24)
Drug: Standard treatment of Covid-19 — Patients will be given Standard treatment of Covid-19 which accordance with National protocol

SUMMARY:
In this randomized controlled trial (RCT), severe cases of COVID-19 infection will be treated with secretome of hypoxia-mesenchymal stem cells. The improvement in clinical, laboratory, and radiological manifestations will be evaluated in treated patients compared with the control group.

DETAILED DESCRIPTION:
The devastating effect of severe acute respiratory syndrome coronavirus-2 (SARS COV-2) infection is caused by a robust cytokine storm that leads to lung tissue damage. Several studies reported a correlation between disease severity and the release of excessive proinflammatory cytokines, such as tumor necrosis factor-α (TNF-α), IL-6, IL-1, IFN-Υ, IFN-Υ-induced protein 10 (IP10), monocyte chemoattractant protein-1 (MCP-1), macrophage inflammatory protein-1a (MIP-1a), and granulocyte-colony stimulating factor (G-CSF). This finding was confirmed by the high level of plasma cytokines found in most severe COVID-19 patients associated with extensive lung damage. Therefore, finding an effective therapeutic option to control the devastating cytokine storm of COVID-19 and regenerate the damaged lung is crucial.

Previous studies reported that the hypoxic condition of MSCs could enhance the release of their active soluble molecules known as Secretome-MSCs (S-MSCs), such as IL-10 and TGF-β that useful in alleviating inflammation. Moreover, they could also increase the expression of growth factors such as VEGF and PDGF that accelerate lung injury improvement. These active molecules could potentially serve as a biological therapeutic agent for treating the severe SARS-CoV-2 infection. According to recent studies, we successfully isolated the S-MSCs from their culture medium using tangential flow filtration (TFF) strategy with several molecular weight cut-off category. This study investigated the clinical outcomes of severe COVID-19 patients with several comorbidities treated with S-MSCs in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose clinical and laboratory test results have a positive diagnosis of Covid-19.
2. Patients who are willing to participate as subjects in the study by signing the informed content.
3. Criteria for Berlin to enter ARDS (moderate and severe) with or without a ventilator:

   * PaO2 / FiO2: moderate 100-200
   * PaO2 / FiO2: severe <100
4. One or more comorbid history
5. SOFA score

Exclusion Criteria:

1. The Covid19 patient has fibrosis (based on the results of the chest X-ray or CT chest)
2. ECOG 4 performance status, decreased irreversible consciousness, brain stem death.
3. Severe NYHA III / IV heart failure
4. Pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in patients clinical manifestation | 1 months
  mild, moderate, or severe
Need for a ventilator | 1 months
  There are respiratory variables that made severe Covid-19 patients previously stable but worsened, requiring a ventilator
  Divided into two categories:
  1. It is necessary
  2. No need
Duration of using a ventilator | 1 months
  Duration of use of a ventilator from the day of intubation to the day of extubation
Length of stay | 1 months
  The length of stay from the first treatment to the patient's final outcome, recovery, or death
Routine blood profile | 2 weeks
  Obtained from patients before and after treatment
CRP | 2 weeks
  Obtained from patients before and after treatment
D-dimer | 2 weeks
  Obtained from patients before and after treatment
Blood Gas Analisis (BGA) | 2 weeks
  Obtained from patients before and after treatment
Photo thorax | 2 weeks
  Obtained from patients before and after treatment

SECONDARY OUTCOMES:
Survival | 2 months
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Agung Putra, Assoc.Prof, Principal Investigator — Stem Cell and Cancer Research Indonesia
Locations (6):
- Indonesia (6):
  - RSUD Bantul, Bantul, Central Java
  - RS PKU Muhammadiyah Gamping, Yogyakarta, Central Java
  - RS Primaya Bekasi Timur, Bekasi, Jakarta Special Capital Region
  - Bhayangkara Hospital, Makassar, South Celebes
  - Gatot Soebroto Army Hospital, Jakarta
  - Dr. Esnawan Antariksa Air Force Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Chen L, Xu Y, Zhao J, Zhang Z, Yang R, Xie J, Liu X, Qi S. Conditioned medium from hypoxic bone marrow-derived mesenchymal stem cells enhances wound healing in mice. PLoS One. 2014 Apr 29;9(4):e96161. doi: 10.1371/journal.pone.0096161. eCollection 2014. PMID 24781370
- [Background] Haraszti RA, Miller R, Stoppato M, Sere YY, Coles A, Didiot MC, Wollacott R, Sapp E, Dubuke ML, Li X, Shaffer SA, DiFiglia M, Wang Y, Aronin N, Khvorova A. Exosomes Produced from 3D Cultures of MSCs by Tangential Flow Filtration Show Higher Yield and Improved Activity. Mol Ther. 2018 Dec 5;26(12):2838-2847. doi: 10.1016/j.ymthe.2018.09.015. Epub 2018 Sep 22. PMID 30341012
- [Result] Harrell CR, Jovicic BP, Djonov V, Volarevic V. Therapeutic Potential of Mesenchymal Stem Cells and Their Secretome in the Treatment of SARS-CoV-2-Induced Acute Respiratory Distress Syndrome. Anal Cell Pathol (Amst). 2020 Nov 20;2020:1939768. doi: 10.1155/2020/1939768. eCollection 2020. PMID 33274176
- [Result] Johnson BS, Laloraya M. A cytokine super cyclone in COVID-19 patients with risk factors: the therapeutic potential of BCG immunization. Cytokine Growth Factor Rev. 2020 Aug;54:32-42. doi: 10.1016/j.cytogfr.2020.06.014. Epub 2020 Jul 1. PMID 32747157